CLINICAL TRIAL: NCT04866394
Title: Stereotactic Pelvic Adjuvant Radiation TherApy in Cancers of the UteruS): A Phase I/II Study (SPARTACUS)
Brief Title: Stereotactic Pelvic Adjuvant Radiation TherApy in Cancers of the UteruS
Acronym: SPARTACUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Eric Leung, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPARTACUS
Record Dates: First submitted 2019-05-14; First posted 2021-04-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: It's a Phase I feasibility study, 5 fractions (hypofractionation)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypofractionated Pelvic Radiation (Experimental)
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Patients will be planned with the aim of delivering 30 Gy in 5 fractions.

SUMMARY:
Advanced technology has enabled radiation oncologists to more accurately and precisely target radiation to areas at risk while maximally sparing healthy tissue. A secondary result of these technologic advances has been the increased utilization of hypofractionationed treatment protocols, since the combined ability to better visualize and precisely deliver radiation to target volumes has allowed radiation oncologists to leverage the therapeutic ratio toward higher target doses whilst maintaining safe doses to the pertinent organs-at-risk. The spectrum of hypofractionation ranges from what are considered moderate (ie. 2- 5 Gy / fraction) into the realm of what is more commonly referred to as stereotactic body (SBRT), generally >5 Gy / fraction. There is growing evidence demonstrating both safety and efficacy for SBRT. The investigators propose that these advantages are translatable to the adjuvant treatment of endometrial cancer.

The investigators submit that a prescription dose of 30 Gy in 5 fractions. Through precision delivery and careful dosimetry the treatment should be safe and well tolerated with minimal impact on patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed endometrial adenocarcinoma
* Patient is a candidate for adjuvant pelvic radiation (+/- vault brachytherapy), meeting one of the following conditions:

  * Patient has serous, clear cell, carcinosarcoma or differentiated histologies.
  * Outer-half myometrial invasion and FIGO grade 1-2 OR
  * FIGO stage II - IIIC1.
* Willing and able to give informed consent to participate in this clinical trial.
* Age ≥18 years.
* Are to receive adjuvant systemic therapy in addition to pelvic radiotherapy will be eligible provided that there is at minimum a 3-week interval between any radiation treatment and chemotherapy treatments.
* Willing and able to complete the QLQ-C30 questionnaire with EN-24 companion as described in the study protocol.
* Primary language of the patient must be English or, if a patient's primary language is not English, they are still able to participate provided the QLQ-C30 and EN-24 is available in their primary language.

Exclusion Criteria:

* Has had prior pelvic radiotherapy.
* Has a contraindication to pelvic radiotherapy, such as but not limited to a connective tissue disease or inflammatory bowel disease.
* Has a contraindication to iodinated CT contrast.
* Has a hip prosthesis.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Acute toxicities | Baseline to 12 weeks following RT completion
  To assess the acute urinary and bowel toxicities associated with adjuvant SBRT treatment in the setting of high-risk endometrial cancer using CTCAE.

SECONDARY OUTCOMES:
Quality of life through EORTC QLQ-C30 and EN24 | Study activation through 2 years post-RT
  To assess the effect of adjuvant SBRT treatment on acute and late patient reported health quality of life using EORTC questionnaires.
Late toxicities | 12 weeks post-RT to 2 years post-RT
  To assess the late urinary, bowel, and other toxicities associated with adjuvant SBRT treatment in the setting of high-risk endometrial cancer using CTCAE.
Local-regional failure | Study activation through 2 years post-RT
  To assess the local-regional failure of adjuvant SBRT treatment by observation of progression or persistence of disease.
Disease-free survival | Study activation through 2 years post-RT
  To document the disease-free survival of those treated with adjuvant SBRT
Dosimetric feasibility | Baseline to RT completion
  The number of patients eligible for enrollment at a 30Gy prescription dose based rigid dosimetric constraints, as compared to a 27.5 Gy treatment dose.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Leung, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung E, Gladwish AP, Davidson M, Taggar A, Velker V, Barnes E, Mendez L, Donovan E, Gien LT, Covens A, Vicus D, Kupets R, MacKay H, Han K, Cheung P, Zhang L, Loblaw A, D'Souza DP. Quality-of-Life Outcomes and Toxic Effects Among Patients With Cancers of the Uterus Treated With Stereotactic Pelvic Adjuvant Radiation Therapy: The SPARTACUS Phase 1/2 Nonrandomized Controlled Trial. JAMA Oncol. 2022 Jun 1;8(6):1-9. doi: 10.1001/jamaoncol.2022.0362. PMID 35420695